CLINICAL TRIAL: NCT06655948
Title: Outcome-related Performance Evaluation Through Revision and Analysis of inTraoperative Events
Acronym: OPERATE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6456
Record Dates: First submitted 2024-09-27; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Laparoscopic Abdominal Surgery
Keywords: Intraoperative Adverse Events; Video-Based Assessment; Minimally Invasive Surgery; Surgical Performance; Patient Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective, multicentric, observational, cohort study is to evaluate intraoperative adverse events (iAEs) through video-based assessment (VBA) across minimal invasive procedures performed in general surgery departments. The main questions it aims to answer are:

* The prevalence, type, and severity of iAEs
* Correlation between iAE and clinical outcomes
* Correlation between iAE and surgical performance
* Qualitative analysis of root cause analysis and mitigation strategies

DETAILED DESCRIPTION:
The OPERATE study is a prospective, multicenter observational cohort study focused on evaluating the prevalence and impact of intraoperative adverse events (iAEs) during minimally invasive surgeries. The study aims to systematically collect and analyze surgical videos and clinical outcomes from multiple centers. By using advanced video-based assessment (VBA) tools, such as the Objective Clinical Human Reliability Analysis (OCHRA) and the Severity of Intraoperative Events and Rectification (SEVERE) index, the study will examine how surgical performance correlates with post-operative outcomes.

The study will initially focus on colorectal surgery, with the possibility of expanding to other types of minimally invasive procedures. Videos of the surgeries will be recorded, de-identified, and uploaded to a centralized platform for analysis. The study also seeks to identify root causes of iAEs and develop strategies to prevent them. Data collection will include not only video-based assessments but also patient demographic details, surgical history, and post-operative recovery data.

By understanding the frequency and nature of iAEs, this study aims to improve surgical safety, reduce complications, and ultimately enhance the quality of patient care in a broad range of general surgical procedures. The findings may contribute to developing new training protocols, artificial intelligence instruments to model errors and increase procedural safety, and guidelines to optimize surgical performance and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective minimally-invasive surgery in participating centers
* Patients with no contraindication to anesthesia and laparoscopic procedures
* Capable of providing informed consent

Exclusion Criteria:

* Surgery performed with palliative intent or under unplanned/emergency setting
* Pregnant or breastfeeding patient
* Patient under legal custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting eligibility criteria and scheduled for elective minimally-invasive surgery in the general surgery departments of participating centers.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intraoperative adverse events | Day of the surgical procedure (1 day)
  The prevalence of iAEs will be assessed using validated VBA tools including the Objective Clinical Human Reliability Analysis (OCHRA), the European Association for Endoscopic Surgery (EAES) classification, and the Severity of Intraoperative Events and Rectification (SEVERE) index.

SECONDARY OUTCOMES:
Outcomes correlation | From the day of the surgical procedure up to 5 years of follow up
  Correlation between iAE and clinical outcomes, overall and per iAEs severity
Severity | Day of the surgical procedure (1 day)
  Prevalence per severity of iAE
Video-Based Assessment | Day of the surgical procedure (1 day)
  Correlation between iAE and surgical performance assessed through validated VBA tools
Root causes | Day of the surgical procedure (1 day)
  Qualitative analysis of root cause analysis and mitigation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Alfieri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (5):
- IHU Strasbourg, Strasbourg, France
- Italy (4):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Isola TIberina - Gemelli Isola, Rome, RM
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RO